CLINICAL TRIAL: NCT07361718
Title: Comparison Between Two Medical Devices for the Reconditioning of Lung Grafts: Pilot Study EVOLUTION (Ex viVO Lung perfUsion for Lung Transplantation)
Brief Title: Comparison Between Two Medical Devices for the Reconditioning of Lungs Intended for Transplantation
Acronym: EVOLUTION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Filippo Antonacci, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 697/2024/Disp/AOUBo
Record Dates: First submitted 2025-11-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Lung Transplant Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCS (Experimental)
  Interventions: Device: Organ Care system
- X vivo (Experimental)
  Interventions: Device: ex vivo lung perfusion for eventual lung transplant

INTERVENTIONS:
Device: ex vivo lung perfusion for eventual lung transplant — ex vivo lung repefusion to evaluate lung function
  Arms: X vivo
Device: Organ Care system — organ care system
  Arms: OCS

SUMMARY:
This study aims to evaluate the effectiveness of two medical devices ( XPS XVIVO and OCS Transmedics) used for organ reperfusion in patients needing bilateral lung transplants from marginal donors.

DETAILED DESCRIPTION:
Marginal organs, which do not have ideal transplant characteristics but are not rejected, can be treated with ex-vivo reperfusion and reventilation machines to optimize their condition. The two main devices studied are:

Organ Care System (OCS) Transmedics, a mobile machine for use at the donor site.

XPS XVIVO, a static machine used for organs transported with cold preservation. The study's primary objective is to assess the acceptance rate of organs treated with these devices, while secondary objectives include comparing the duration of mechanical ventilation, ECMO use, and 90-day survival rates in transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* informed consent
* donor with at least one of the following: age greater than 55 years P/F on evaluation less than 350 mmHg smoker (more than 20 p/y) lung atelectasis on chest ct class II and III DCD according to Maastricht classification

Exclusion Criteria:

* lung Haematoma or signsd of lung contusion
* signs of infecton of the graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptance rate to transplant | after the transplant

SECONDARY OUTCOMES:
days on mechanical ventilation | from transplant moment since the day weaning from mechanical ventilation
duration on postoperative ECMO (ExtraCorporeal Membrane Oxygenation) | from transplant date since the day weaning from ECMO (ExtraCorporeal Membrane Oxygenation)
mortality | within 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Aoubo, Bologna, BO, Italy